CLINICAL TRIAL: NCT00467337
Title: Medial-Wedge Insole is Highly Effective in the Treatment of Valgus Knee Osteoarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPPESP#130/04
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Osteoathritis
Keywords: insole; osteoarthritis; pain; valgus knee
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Medial-Wedge Insole intervention

SUMMARY:
* To assess the efficacy of medial-wedge insole in valgus knee osteoarthritis (OA).
* We hypothesized that medial-wedged insoles are biomechanically effective and should reduce lateral compartment loading in persons with valgus knee osteoarthritis with a consequent symptomatic improvement.

DETAILED DESCRIPTION:
Thirty females fulfilling the American College of Rheumatology criteria for knee osteoarthritis with bilateral valgus deformity greater than or equal to 8° were consecutively will be selected from the Rheumatology Outpatient Clinic of University of São Paulo. Radiographic grading of OA was defined according to Kellgren and Lawrence (KL) and analyzed blind by the same rheumatologist. Inclusion criteria were knee osteoarthritis with lateral compartment involvement detected on X-Ray (KL class II or more); absence or minimal (KL class 0 or I) for medial compartment involvement; and pain on movement > 2 measured by Visual Analog Scale (VAS).

Exclusion criteria were: body mass index (BMI) > 40, scoliosis, lower limbs length difference exceeding 1 cm, knee surgery, hallux rigidus, previous history of rheumatologic disease (rheumatoid arthritis, connective tissue disease, microcrystalline arthropathy, and soronegative arthropathy), soft tissue involvement (anserine, patellar, and calcaneal tendinopathy), and foot/lower leg symptoms.

Corticosteroid and hyaluronic acid infiltrations were not allowed 3 and 6 months prior to entry, respectively. The use of non-steroidal anti-inflammatory and analgesics or slow action drugs (DMARDs) were allowed if prescribed at least four weeks and eight weeks before entry and remained unchanged throughout the study.

The study was approved by the local Ethical Committee and all patients signed informed consent.

Study protocol:

Patients will be randomly assigned into 2 groups: CASES with 16 patients and CONTROLS with fourteen patients. The CASES wore 8 mm high, medial-wedged insoles for the hind foot inserted into a new shoe for 8 weeks. The CONTROLS will use an insole resembling the former group, only without raised wedges (FIGURE 1-B) for 8 weeks. Patients of both groups will receive the same new shoe and were blind to the insole use.

The ethylene-vinyl-acetate (EVA - density 50) insoles were provided by the AACD Institute (Handicapped Child Care Association). A commercial neoprene with elastic banding will be used for ankle support. Both groups will use similar standard shoes supplied by the hospital. Each participant will be instructed to use the splints (shoes and elastic banding) for 3 to 6 hours daily. The correct use of the splints will be checked every two weeks. Undesirable side-effects will be recorded at the end of the study.

Age, disease duration, weight, height, body mass index (BMI), and sedentarism (only daily activities) will be recorded for all patients at entry. In order to assess symptoms, Visual Analog Scale (VAS) will be used for night pain, pain at rest and on movement. Lequesne index score and the WOMAC questionnaire will be applied at baseline and after 8 weeks by a blinded examiner.

Antero-posterior conventional X-ray of knees and ankles will be performed under monopodalic load with and without insoles in order to measure femorotibial, talocalcaneal, and talus tilt angles. Femorotibial angle is formed by the intersection of femur and tibia axes, obtained through lines drawn at distal one-third of the femur and proximal one-third of the tibia, both equidistant from external limits of the cortical bones. Talocalcaneal angle is formed by a first line connecting the midpoints between the trochanter talus to the lateral and medial malleoli, and a second line perpendicular to the floor identified by inferior border of X-ray. Tilt angle of talus is formed by a line parallel to floor and the tilt of the trochanter talus. All angles will be measured blind by the same rheumatologist.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis with bilateral valgus deformity greater than or equal to 8°.
* Radiographic grading of OA was defined according to Kellgren and Lawrence (KL)class II or more
* pain on movement > 2 measured by Visual Analog Scale (VAS).

Exclusion Criteria:

* body mass index (BMI) > 40
* scoliosis
* lower limbs length difference exceeding 1 cm
* knee surgery
* hallux rigidus
* previous history of rheumatologic disease (rheumatoid arthritis, connective tissue disease, microcrystalline arthropathy,soronegative arthropathy)
* soft tissue involvement (anserine, patellar, and calcaneal tendinopathy)
* foot/lower leg symptoms

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To assess symptoms, Visual Analog Scale (VAS) will be used for night pain, pain at rest and on movement. Lequesne index score and the WOMAC questionnaire will be applied at baseline and after 8 weeks by a blinded examiner. | 2 years

SECONDARY OUTCOMES:
Antero-posterior conventional X-ray of knees and ankles were both performed under monopodalic load with and without insoles in order to measure femorotibial, talocalcaneal, and talus tilt angles. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Fuller, MD PhD, Principal Investigator — Rheumatology Division HCFMUSP; Eloisa Bonfa, MD PhD, Study Director — Rheumatology Division HCFMUSP

REFERENCES:
- [Derived] Rodrigues PT, Ferreira AF, Pereira RM, Bonfa E, Borba EF, Fuller R. Effectiveness of medial-wedge insole treatment for valgus knee osteoarthritis. Arthritis Rheum. 2008 May 15;59(5):603-8. doi: 10.1002/art.23560. PMID 18438931